CLINICAL TRIAL: NCT04622644
Title: A Pilot Study Using a Microwave Device for Stroke Detection (StrokeWave) to Discriminate Between Haemorragic and Ischaemic Stroke
Brief Title: Clinical Investigation to Evaluate the Suitability of StrokeWave in Distinguishing Haemorragic From Ischaemic Strokes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umbria Bioengineering Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UBT-01-20
Record Dates: First submitted 2020-11-02; First posted 2020-11-10 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): All patients perform StrokeWave exam, after NCCT and before CTA acquisition.
  Interventions: Device: Device: clinical investigation microwave device class IIa not marked CE for stroke detection

INTERVENTIONS:
Device: Device: clinical investigation microwave device class IIa not marked CE for stroke detection — Patients with hyperacute stroke are referred to the emergency room with a 'stroke code'. Clinical collected data includes NIHSS and mRS. Patients will undergo to NCCT in order to exclude the haemorragic nature of vascular disease. In the same diagnostic session the patient undergo to CTA with tri-phase protocol to assess LVO. Before starting the CTA acquisition with iodinate contrast injection the StrokeWave will be placed on the head of the patients in the CT room passing toward the gantry of the CT avoiding any loose of time. The scanning with the StrokeWave will be performed in about 5 minutes and the system will be removed allowing the CTA acquisition.

SUMMARY:
This is a pilot, monocentric clinical investigation to evaluate the suitability of StrokeWave in distinguishing haemorragic from ischaemic strokes. The StrokeWave is a microwave device which employs a novel technique to generate images by processing very low power (<1mW) microwaves. The trial design has been developed in order not to interfere with thw standard diagnostic approach used for the hyperacute stroke patients, nor to modify the usual standard timing of the routine assessment.

DETAILED DESCRIPTION:
The number of participants will be 60. Patients with hyperacute stroke (within 4 hours from the onset) or with awake or unknow time of onset strokes will be enrolled in the study. All patients will be registered at emergency room of Hospital, and according to the internal procedure will be clinically evaluated by the Neurologist of the stroke team. NIHSS and mRS will be administered and scores registered. The scanning with StrokeWave will be performed in 5 minutes, after NCCT and before the CTA acquisition, in the CT room. StrokeWave will be placed on the head of the patients in the CT room passing toward the gantry of the CT avoiding any loose of time. After the StrokeWave scanning, the system will be removed. The data collected will be processed through an imaging algorithm which is integrated in the device. The final output will be composed by one or more images, plus one or more parameters describing the images.

ELIGIBILITY:
Inclusion Criteria:

* Adult > 18 years old
* Patients with hyperacute stroke, i.e. which are referred to the emergency room with a 'stroke code'

Exclusion Criteria:

* mRS >3 before the stroke onset
* Life expectancy <3 months
* GCS=3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
To generate empirical evidence that StrokeWave can detect and distinguish beteween haemorragic and ischaemic stroke at the same extent as NCCT | During the baseline
  StrokeWave ability to distinguish between haemorragic and ischaemic stroke compared to NCCT results (concordance between ischaemic and haemorragic strokes identified with 2 methods)

SECONDARY OUTCOMES:
StrokeWave sensitivity in the ischaemic stroke | During the baseline
  To measure the sensitivity of StrokeWave in the ischaemic stroke (ASPECT scale)
StrokeWave sensitivity in the haemorragic stroke | During the baseline
  To measure the sensitivity of StrokeWave in the haemorragic stroke (site, dimension)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Nuovo Santa Chiara, Pisa, Italy